CLINICAL TRIAL: NCT05386303
Title: Quantitative Pupillometry During External Ventricular Drain Weaning - An Observational Study
Brief Title: Quantitative Pupillometry
Acronym: HYDRO-NiP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC21_0078
Record Dates: First submitted 2021-05-19; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2021-05

CONDITIONS: Hydrocephalus; Critical Care
Keywords: Pupillometry; External ventricular drain; Weaning; Brain injury; Pupillary reactivity
MeSH Terms: conditions — Hydrocephalus; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the diagnostic ability of quantitative pupillometry for the early detection of hydrocephalus during the weaning process of the external ventricular drain.

DETAILED DESCRIPTION:
Acute hydrocephalus is an emergency often requiring the insertion of an external ventricular drain (EVD). In the aftermath, the patient is transferred to an intensive care unit (ICU) for close monitoring. Ensuring optimal cerebral perfusion through efficient drainage of cerebrospinal fluid while minimizing drainage duration are the objectives of care.

Assessing pupillary light reflex is a key test for the detection of neurological deterioration. For long, this assessment has been grossly performed via a qualitative approach (present/absence of pupillary light reflex). For a more precise assessment, quantitative pupillometry has been proposed. Pupil size and constriction speed in response to a standard light are recorded by an automatic portable and user-friendly device. This device is increasingly used in the ICU, mostly for prognostication after acute brain injury. We hypothesized that quantitative pupillometry parameters may vary when hydrocephalus occurs.

The aim of this study is to assess whether quantitative pupillometry parameters vary when hydrocephalus occurs. The investigators focused on the early detection of hydrocephalus during the EVD weaning process.

ELIGIBILITY:
Inclusion Criteria :

* Patient older than 18 years old
* Admitted to the ICU
* With an external ventricular drain
* Consenting to participate (or consent from his/her next of kin, if unable to consent).

Exclusion Criteria :

* Patient with pre-existing bilateral pupillary pathology
* Pregnant or breast-feeding patient
* Moribund patient or patient with decision of withholding or withdrawing life-sustaining treatment
* Patient with no health insurance
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients with an EVD included at the beginning of the weaning process
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-31 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
NPi (Neurological Pupil index) and EVD (external ventricular drain)occlusion test | 5 days
  NPi will be compared between two groups of patients (constituted a posteriori): success and failure of the EVD occlusion test.
  Independently of this study, the EDV occlusion test starts as soon as prescribed by the physician as a prerequisite before its withdrawal.
  Failing an occlusion test is defined by the need for reopening the EVD.

SECONDARY OUTCOMES:
Diagnostic evaluation | 5 days
  Pupillometer ability to detect an EDV occlusion test failure will be studied. The area under the ROC curve (AUCROC) will be determined. We define, a priori, that the detection performance will be, respectively, honorable, good or excellent if the AUCROC is higher than 0.70, 0.80 and 0.90.
Pupillometry and EVD occlusion test | 5 days
  Constriction velocity will be compared between two groups of patients (constituted a posteriori): success and failure of the occlusion test.
Dilatation velocity | 5 days
  Dilation velocity will be compared between two groups of patients (constituted a posteriori): success and failure of the occlusion test.
Maximum constriction velocity | 5 days
  Maximum constriction velocity will be compared between two groups of patients (constituted a posteriori): success and failure of the occlusion test.
Latency of contraction | 5 days
  Latency of contraction will be compared between two groups of patients (constituted a posteriori): success and failure of the occlusion test.
Pupil size variation | 5 days
  Pupil size variation will be compared between two groups of patients (constituted a posteriori): success and failure of the occlusion test.
Pupillometry and clinical scores | 5 days
  The association between pupillometry parameters and clinical scores (Glasgow Coma Scale, FOUR score, RASS and CAM-ICU) will be studied
The association between pupillometry parameters and ventricular volume will be studied. | 5 days
  A relationship between, measurements of ventricular volumes (via brain imaging examinations performed regardless of this study) and pupillometry parameters will be sought

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme DAUVERGNE, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - Nantes University Hospital, Nant, Loire-Atlantique
  - CHU de Nantes, Nantes

IPD SHARING:
Plan to Share IPD: Undecided